CLINICAL TRIAL: NCT02550405
Title: The Behavioral and Brain Mechanism of Internet Gaming Disorder
Brief Title: The Behavioral and Brain Mechanism of IGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, jintao, zhang, Associated Professor, Beijing Normal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeijingNormalU
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Craving behavioral intervention (Experimental): The craving behavioral intervention (CBI) was developed based on the framework of craving, combining with behavior intervention (Dong and Potenza, 2014), and conducted among individuals with IGD.
  Interventions: Behavioral: Craving behavioral intervention
- Control (No Intervention): The control group were individuals with Internet gaming disorder who did not receive any intervention but were scanned twice with the similar interval period as experimental group.

INTERVENTIONS:
Behavioral: Craving behavioral intervention — The CBI was given once a week for 6 weeks, conducted by four therapists. A pair of therapists was randomly assigned to a CBI+ group. Each session included 5 parts in 2.5-3 hours: warming-up exercise, discussion about the homework from the last session, main structured activity, brief summary, and the homework assignment. There were 6 sessions with each focused on a topic: recognize craving and its relationship with IGD; reduce craving through ameliorating the salience of cues and irrational beliefs, withdrawal symptoms and other negative affects; enhance self-monitoring and control for craving through time management training; relieve fulﬁllment of psychological needs through Internet use and attenuate the relation between craving and gaming behaviors through coping skill training
  Other Names: CBI
  Arms: Craving behavioral intervention

SUMMARY:
This project aims to investigate whether anodal tDCS of dlPFC enhances cognitive regulation over craving an emotions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for IGDs were:

  1. a score of 67 or higher on the CIAS;
  2. engagement in Internet gaming for over 14 hours per week for a minimum of one year; and
  3. reporting of Internet gaming as their primary online activity;
* Inclusion criteria for HCs were:

  1. a score < 60 on the CIAS;
  2. never having spent more than 2 hours per week engaged in Internet gaming

Exclusion Criteria:

* for all participants:

  1. current or history of use of illegal substances and gambling;
  2. current or history of psychiatric or neurological illness; and
  3. current use of psychotropic medications

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Brain resting state functional connectivity as measured by fMRI | Detecting changes between two different time points (baseline and 6 weeks)
  voxel-wise, ROI-wise, and ICA analyses
Brain activation during a cue-induced craving task as measured by fMRI | Detecting changes between two different time points (baseline and 6 weeks)
  A paradigm using addictive pictures to induce craving

SECONDARY OUTCOMES:
Brain activation during the Cups task as measured by fMRI | Detecting changes between two different time points (baseline and 6 weeks)
  Cups task measuring risky decision-making related to potential gains and losses separately
Brain activation during the mixed gambling task tasks as measured by fMRI | Detecting changes between two different time points (baseline and 6 weeks)
  The mix gambling task measuring decision-making related to loss aversion
Brain structure as measured by structural MRI | Detecting changes between two different time points (baseline and 6 weeks)
  comparing gray matter and white matter differences between individuals with IGD and healthy controls.
IGD severity measured by Chen Internet addiction scale | Detecting changes between two different time points (baseline and 6 weeks)
  a 26-item 4-point Likert scale
Craving as measured by brief questionnaire of Internet (gaming) craving | Detecting changes between two different time points (baseline and 6 weeks)
  a 8-item 7-point Likert scale
Impulsivity as measured by Barratt impulsive scale (BIS-II) | Detecting changes between two different time points (baseline and 6 weeks)
  a 30-item 4-point Likert scale
weekly online (gaming) time | Detecting changes between two different time points (baseline and 6 weeks)
  self-report,in hours

CONTACTS AND LOCATIONS:
Overall Officials: XiaoYi Fang, PhD, Study Chair — Institute of Developmental Psychology, Beijing Normal University; JinTao Zhang, PhD, Study Chair — State Key Laboratory of Cognitive Neuroscience and Learning; CuiCui Xia, MEd, Principal Investigator — Institute of Developmental Psychology, Beijing Normal University; LinYuan Deng, PhD, Principal Investigator — Faculty of Education Beijing Normal University; Lu Liu, BS, Principal Investigator — Institute of Developmental Psychology, Beijing Normal University; Ben Liu, BSM, Principal Investigator — State Key Laboratory of Cognitive Neuroscience and Learning; ShanShan Ma, BS, Principal Investigator — State Key Laboratory of Cognitive Neuroscience and Learning; YuanWei Yao, BS, Principal Investigator — State Key Laboratory of Cognitive Neuroscience and Learning; Qinxue Liu, PhD, Principal Investigator — School of Psychology Central China Normal University; Nan Zhou, MEd, Principal Investigator — Institute of Developmental Psychology, Beijing Normal University; ShuMeng Hou, MEd, Principal Investigator — Institute of Developmental Psychology, Beijing Normal University
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Dong G, Potenza MN. A cognitive-behavioral model of Internet gaming disorder: theoretical underpinnings and clinical implications. J Psychiatr Res. 2014 Nov;58:7-11. doi: 10.1016/j.jpsychires.2014.07.005. Epub 2014 Jul 17. PMID 25062755
- [Derived] Liu L, Yao YW, Li CR, Zhang JT, Xia CC, Lan J, Ma SS, Zhou N, Fang XY. The Comorbidity Between Internet Gaming Disorder and Depression: Interrelationship and Neural Mechanisms. Front Psychiatry. 2018 Apr 23;9:154. doi: 10.3389/fpsyt.2018.00154. eCollection 2018. PMID 29740358
- [Derived] Deng LY, Liu L, Xia CC, Lan J, Zhang JT, Fang XY. Craving Behavior Intervention in Ameliorating College Students' Internet Game Disorder: A Longitudinal Study. Front Psychol. 2017 Apr 10;8:526. doi: 10.3389/fpsyg.2017.00526. eCollection 2017. PMID 28443046